CLINICAL TRIAL: NCT02519972
Title: Low-dose Computed Tomography Screening for Lung Cancer in Relatives With Family History of Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuo-Husan Hsu, Attending physician, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: DOH96-TD-G-111-016
Record Dates: First submitted 2015-07-31; First posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Lung Cancer
Keywords: Low dose CT screening; Family history of lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Low dose computed tomography (Experimental): All the Low dose computed tomography of lung was performed with 64 slices multidetectors CT in single hold breath covering entire lung. The protocol of scanning parameters (120KVp, 40-80 mA, 1.25 mm or less in thickness) was standardized. The raw data would be reconstructed to axial images (3 mm thickness and interval) and coronal images (3 mm thickness and interval). The scan should be finished in a single breath (15-20 second) from the thoracic inlet to adrenal glands.
  Interventions: Device: low dose computed tomography

INTERVENTIONS:
Device: low dose computed tomography — Participants will receive 3 round of low dose computed tomography screening every year

SUMMARY:
Screening with the use of low-dose computed tomography (LDCT) reduces mortality from lung cancer. Relatives with family history of lung cancer are at increased risk of lung cancer compared to those without a family history in pooled analysis. A prospective trial using LDCT of lung to screen the relatives with family history of lung cancer is needed.

DETAILED DESCRIPTION:
Investigators invited participants with family history to join in this study under the criteria of (1) relatives of the lung cancer patients; (2) age older than 55 years old or age older than the age of onset of lung cancer proband if the family members were less than 55 years old; (3) compulsory signing the consent agreement after understanding the purpose of study and the exposure of radiation. The participants with (1) proved lung cancer either with or without treatment, (2) presence of hemoptysis or history of remarkable lung fibrosis, (3) any other cancer history or (4) chest CT examination within one year would be excluded from the study.

The study was planned to enroll 1000 participants from simplex families and 500 participants from multiplex families for lung LDCT screening. Multiplex family was defined as two or more family members with lung cancers, and simplex family as one family member with lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. relatives of the lung cancer patients;
2. age older than 55 years old or age older than the age of onset of lung cancer proband if the family members were less than 55 years old;
3. compulsory signing the consent agreement after understanding the purpose of study and the exposure of radiation.

Exclusion Criteria:

1. proved lung cancer either with or without treatment,
2. presence of hemoptysis or history of remarkable lung fibrosis,
3. any other cancer history or
4. chest CT examination within one year

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1102 (Actual)
Dates: Start 2007-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with lung cancer detected by low dose computed tomography | three years

SECONDARY OUTCOMES:
Detection rate of early lung cancer | three years

CONTACTS AND LOCATIONS:
Overall Officials: Gee-Chen Chang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital

REFERENCES:
- [Background] Sun S, Schiller JH, Gazdar AF. Lung cancer in never smokers--a different disease. Nat Rev Cancer. 2007 Oct;7(10):778-90. doi: 10.1038/nrc2190. PMID 17882278
- [Background] Katanoda K, Marugame T, Saika K, Satoh H, Tajima K, Suzuki T, Tamakoshi A, Tsugane S, Sobue T. Population attributable fraction of mortality associated with tobacco smoking in Japan: a pooled analysis of three large-scale cohort studies. J Epidemiol. 2008;18(6):251-64. doi: 10.2188/jea.je2007429. Epub 2008 Dec 9. PMID 19075498
- [Background] Chen CJ, Wu HY, Chuang YC, Chang AS, Luh KT, Chao HH, Chen KY, Chen SG, Lai GM, Huang HH, et al. Epidemiologic characteristics and multiple risk factors of lung cancer in Taiwan. Anticancer Res. 1990 Jul-Aug;10(4):971-6. PMID 2382996
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Sone S, Takashima S, Li F, Yang Z, Honda T, Maruyama Y, Hasegawa M, Yamanda T, Kubo K, Hanamura K, Asakura K. Mass screening for lung cancer with mobile spiral computed tomography scanner. Lancet. 1998 Apr 25;351(9111):1242-5. doi: 10.1016/S0140-6736(97)08229-9. PMID 9643744
- [Background] Matakidou A, Eisen T, Houlston RS. Systematic review of the relationship between family history and lung cancer risk. Br J Cancer. 2005 Oct 3;93(7):825-33. doi: 10.1038/sj.bjc.6602769. PMID 16160696
- [Background] Cote ML, Liu M, Bonassi S, Neri M, Schwartz AG, Christiani DC, Spitz MR, Muscat JE, Rennert G, Aben KK, Andrew AS, Bencko V, Bickeboller H, Boffetta P, Brennan P, Brenner H, Duell EJ, Fabianova E, Field JK, Foretova L, Friis S, Harris CC, Holcatova I, Hong YC, Isla D, Janout V, Kiemeney LA, Kiyohara C, Lan Q, Lazarus P, Lissowska J, Le Marchand L, Mates D, Matsuo K, Mayordomo JI, McLaughlin JR, Morgenstern H, Mueller H, Orlow I, Park BJ, Pinchev M, Raji OY, Rennert HS, Rudnai P, Seow A, Stucker I, Szeszenia-Dabrowska N, Dawn Teare M, Tjonnelan A, Ugolini D, van der Heijden HF, Wichmann E, Wiencke JK, Woll PJ, Yang P, Zaridze D, Zhang ZF, Etzel CJ, Hung RJ. Increased risk of lung cancer in individuals with a family history of the disease: a pooled analysis from the International Lung Cancer Consortium. Eur J Cancer. 2012 Sep;48(13):1957-68. doi: 10.1016/j.ejca.2012.01.038. Epub 2012 Mar 19. PMID 22436981
- [Background] International Early Lung Cancer Action Program Investigators; Henschke CI, Yankelevitz DF, Libby DM, Pasmantier MW, Smith JP, Miettinen OS. Survival of patients with stage I lung cancer detected on CT screening. N Engl J Med. 2006 Oct 26;355(17):1763-71. doi: 10.1056/NEJMoa060476. PMID 17065637
- [Background] Sone S, Li F, Yang ZG, Honda T, Maruyama Y, Takashima S, Hasegawa M, Kawakami S, Kubo K, Haniuda M, Yamanda T. Results of three-year mass screening programme for lung cancer using mobile low-dose spiral computed tomography scanner. Br J Cancer. 2001 Jan 5;84(1):25-32. doi: 10.1054/bjoc.2000.1531. PMID 11139308
- [Background] Nawa T, Nakagawa T, Kusano S, Kawasaki Y, Sugawara Y, Nakata H. Lung cancer screening using low-dose spiral CT: results of baseline and 1-year follow-up studies. Chest. 2002 Jul;122(1):15-20. doi: 10.1378/chest.122.1.15. PMID 12114333
- [Background] New York Early Lung Cancer Action Project Investigators. CT Screening for lung cancer: diagnoses resulting from the New York Early Lung Cancer Action Project. Radiology. 2007 Apr;243(1):239-49. doi: 10.1148/radiol.2431060467. PMID 17392256